CLINICAL TRIAL: NCT01743729
Title: A Phase 3, Multicenter, Randomized, Double-Masked and Placebo-Controlled Study Evaluating the Efficacy of a 5.0% Concentration of Lifitegrast Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye Currently Using Artificial Tears (OPUS-2)
Brief Title: A Phase 3 Study to Evaluate the Efficacy of Lifitegrast in Subjects With Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1118-DRY-300
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Dry Eye Disease
Keywords: SAR 1118
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifitegrast (Experimental): Lifitegrast Ophthalmic Solution (5.0%)
  Interventions: Drug: Lifitegrast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lifitegrast — Lifitegrast Ophthalmic Solution 5.0%
  Other Names: SAR 1118
  Arms: Lifitegrast
Drug: Placebo — Placebo for Lifitegrast Ophthalmic Solution 5.0%
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of lifitegrast ophthalmic solution compared to placebo in the treatment of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read, sign and date the informed consent and HIPAA documents
* Willing and able to comply with all study procedures
* Be at least 18 years of age
* Patient-reported history of dry eye in both eyes
* A negative urine pregnancy test if female of childbearing potential and must use adequate birth control throughout the study period
* Artificial tear use within the past 30 days

Exclusion Criteria:

* Any ocular condition that, in the opinion of the Investigator, could affect study parameters including, but not limited to, active ocular infection, ocular inflammation, glaucoma, and/or diabetic retinopathy
* Unwilling to avoid wearing contact lenses for 7 days prior to first visit and for the duration of the study
* Any blood donation or significant loss of blood within 56 days of Visit 1
* Any history of immunodeficiency disorder, positive HIV, hepatitis B, C, or evidence of acute active hepatitis A (anti-HAV IgM), or organ or bone marrow transplant.
* Use of any prohibited medications at any time during the study unless otherwise specified
* Any significant illness that could interfere with study parameters
* History of laser assisted in situ keratomileusis (LASIK) or similar type of corneal refractive surgery within 12 months prior to first visit, and/or any other ocular surgical procedure within 12 months prior to first visit; or any scheduled ocular surgical procedure during the study period.
* Known history of alcohol and/or drug abuse
* Subjects with Dry eye secondary to scarring or destruction of conjunctival goblet cells (as with Vitamin A deficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (28):
- United States (28):
  - OPUS-2 Investigational Site, Artesia, California
  - OPUS-2 Investigational Site, Hemet, California
  - OPUS-2 Investigational Site, Lancaster, California
  - OPUS-2 Investigational Site, Mission Hills, California
  - OPUS-2 Investigational Site, Montebello, California
  - OPUS-2 Investigational Site, Newport Beach, California
  - OPUS-2 Investigational Site, Petaluma, California
  - OPUS-2 Investigational SIte, Rancho Cordova, California
  - OPUS-2 Investigational Site, Danbury, Connecticut
  - OPUS-2 Investigational Site, Fort Myers, Florida
  - OPUS-2 Investigational Site, Hoffman Estates, Illinois
  - OPUS-2 Investigational Site, Indianapolis, Indiana
  - OPUS-2 Investigational Site, New Albany, Indiana
  - OPUS-2 Investigational Site, Lexington, Kentucky
  - OPUS-2 Investigational Site, Saint Paul, Minnesota
  - OPUS-2 Investigational Site, Chesterfield, Missouri
  - OPUS-2 Investigational Site, Des Peres, Missouri
  - OPUS-2 Investigational Site, Independence, Missouri
  - OPUS-2 Investigational Site, Kansas City, Missouri
  - OPUS-2 Investigational Site, Washington, Missouri
  - OPUS-2 Investigational Site, New York, New York
  - OPUS-2 Investigational Site, Wantagh, New York
  - OPUS-2 Investigational Site, Cleveland, Ohio
  - OPUS-2 Investigational Site, Philadelphia, Pennsylvania
  - OPUS-2 Investigational Site, Houston, Texas
  - OPUS-2 Investigational Site, League City, Texas
  - OPUS-2 Investigational Site, San Antonio, Texas
  - OPUS-2 Investigational Site, Norfolk, Virginia

REFERENCES:
- [Result] Tauber J, Karpecki P, Latkany R, Luchs J, Martel J, Sall K, Raychaudhuri A, Smith V, Semba CP; OPUS-2 Investigators. Lifitegrast Ophthalmic Solution 5.0% versus Placebo for Treatment of Dry Eye Disease: Results of the Randomized Phase III OPUS-2 Study. Ophthalmology. 2015 Dec;122(12):2423-31. doi: 10.1016/j.ophtha.2015.08.001. Epub 2015 Sep 11. PMID 26365210

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two of 720 participants were excluded from data analysis due to duplication. Therefore, 718 participants were randomized and treated. One participant from placebo arm (N=360) has taken study drug by mistake and considered for "Lifitegrast" arm (N=358). Therefore, Placebo (N=359), Lifitegrast (N=359) were considered for safety analysis.
Period: Overall Study
Arm/Group | Lifitegrast | Placebo
Started | 358 (One participant from placebo arm included in Lifitegrast arm for safety analysis set (N=359).) | 360 (One placebo participant was considered for Lifitegrast arm; Placebo safety analysis set (N= 359).)
Completed | 321 | 348
Not Completed | 37 | 12

BASELINE CHARACTERISTICS:
Population: Randomized population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifitegrast | Placebo | Total
Number analyzed (Participants) | 358 | 360 | 718
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (13.93) | 58.9 (14.26) | 58.8 (14.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 265 | 550
  Male | 73 | 95 | 168

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Inferior Corneal Fluorescein Staining Score to Day 84
Description: Corneal staining was performed to grade the degree of corneal epithelial cell injury as measured by fluorescence using slit-lamp examination. The corneal surface is divided into three regions: superior, central and inferior. The scores for each of these 3 regions ranged from 0 to 4 (0=no staining; 1=few/rare punctate lesions; 2=discrete and countable lesions; 3=lesions too numerous to count, but not coalescent; 4=coalescent) with 0.5 point increments, and lower scores indicate improvement. Inferior corneal fluorescein staining scores from the study eye only were reported. Study eye is the 'worse eye', defined as the eye with worse (higher) score at baseline.
Time Frame: Baseline to Day 84
Population: Intent-to-treat (ITT) set included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast | Placebo
Number analyzed (Participants) | 358 | 360
units on a scale
  Baseline | 2.39 (0.763) | 2.40 (0.722)
  Change from Baseline to Day 84 | -0.73 (0.926) | -0.71 (0.943)
Statistical Analysis 1: Comparison: Lifitegrast vs Placebo; Test type: Superiority or Other; p = 0.6186, ANCOVA; Treatment Effect = 0.03, 95% CI 2-sided [-0.10 to 0.17]

2. Primary Outcome: Change From Baseline in Eye Dryness Score (Visual Analogue Scale) to Day 84
Description: Eye dryness score was assessed on a visual analogue scale (a 7-item [burning/stinging, itching, foreign body sensation, eye discomfort, eye dryness, photophobia, and pain], participant-reported, symptom index) with scores ranging from 0 to 100 (0=no discomfort; 100=maximal discomfort) and lower scores indicate a better outcome.
Time Frame: Baseline to Day 84
Population: ITT population with last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast | Placebo
Number analyzed (Participants) | 358 | 360
units on a scale
  Baseline | 69.68 (16.954) | 69.22 (16.761)
  Change from Baseline to Day 84 | -35.30 (28.400) | -22.75 (28.600)
Statistical Analysis 1: Comparison: Lifitegrast vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Treatment Effect = 12.61, 95% CI 2-sided [8.51 to 16.70]

ADVERSE EVENTS:
Description: One participant from placebo group (N=360) has taken study drug by mistake and considered for "Lifitegrast" group (N=358). Therefore, Placebo (N)= 359, Lifitegrast (N)=359 were considered for safety analysis.
Arm/Group | Lifitegrast | Placebo
Serious Adverse Events (participants affected / at risk) | 3/359 | 4/359
Other Adverse Events (participants affected / at risk) | 102/359 | 30/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifitegrast (N=359) | Placebo (N=359)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyrotoxic crisis (Endocrine disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifitegrast (N=359) | Placebo (N=359)
Visual acuity reduced (Eye disorders) | 18 (23) | 23 (28)
Instillation site irritation (General disorders) | 28 (29) | 5 (5)
Instillation site reaction (General disorders) | 25 (29) | 4 (4)
Dysgeusia (Nervous system disorders) | 58 (58) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicentre publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicentre Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.